CLINICAL TRIAL: NCT05011708
Title: Examining Symptomatic Relief and Kinetic Stability of I-DROP MGD Eye Drops (LIME)
Brief Title: I-DROP MGD Symptomatic Relief and Tear Film Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I-MED Pharma (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDROPMGD072021
Record Dates: First submitted 2021-07-29; First posted 2021-08-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 of the study will be double-masked (both investigator and participant are masked).
  Part 2 will not involve masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (I-DROP MGD) (Experimental): Part I of this study is a contralateral eye design, accordingly patient would receive either I-DROP MGD (Test) or Thealoz Duo (Control) in either eye.
  Part II, patients shall receive either only I-DROP MGD
  Interventions: Device: I-DROP MGD
- Control - Thealoz Duo (Active Comparator): Part I of this study is a contralateral eye design, accordingly patient would receive either I-DROP MGD (Test) or Thealoz Duo (Control) in either eye.
  Part II, patients shall receive either only I-DROP MGD
  Interventions: Device: Thealoz Duo

INTERVENTIONS:
Device: I-DROP MGD — I-DROP MGD are eye drop produced by I-MED PHARMA for the management of moderate to severe Dry Eye Disease.
  Arms: Test (I-DROP MGD)
Device: Thealoz Duo — I-DROP MGD are eye drop produced by Laboratoires Thea for the management of Dry Eye Disease.
  Arms: Control - Thealoz Duo

SUMMARY:
The objective of the study is to compare the difference in tear film stability and symptomatic relief between I-DROP MGD and another commercially available drop in the Canadian market.

DETAILED DESCRIPTION:
The purpose of this study is to:

* Compare tear film measurements for two hours after putting one drop of I-DROP MGD eye drops into one eye and one drop of Thealoz Duo eye drops in the other eye.
* Investigate the relief of dry eye symptoms with I-DROP MGD eye drops after 7 days of use.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Habitually uses ocular lubricants or artificial tears to relieve symptoms of dryness at least once per day for the past 30 days;
5. Has dry eye disease as per the TFOS DEWS II definition:

   1. DEQ-5 ≥ 6 or OSDI ≥ 13
   2. PLUS at least ONE of the following signs in at least one eye:

   i. NITBUT < 10 seconds ii. >5 spots of corneal fluorescein staining OR > 9 conjunctival spots iii. Lid wiper fluorescein staining ≥ 2mm length ≥ 25% width.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has worn any contact lenses in the past 30 days;
3. Has previously, or currently uses I-DROP MGD eye drops;
4. Has any known allergy or intolerance to I-DROP MGD or Thealoz Duo eye drops;
5. Has any known active* ocular disease (allergies or inflammation) and/or infection;
6. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable (e.g. uncontrolled autoimmune disease or uncontrolled immunodeficiency disease);
7. Has a history of sensitivity to rapidly blinking lights or photosensitive epilepsy as one of the a key assessment device employs rapid blinking lights;
8. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable (e.g. antihistamines);
9. Has known sensitivity to sodium fluorescein to be used in the study;
10. Self-reports that they are pregnant, lactating or planning a pregnancy at the time of enrolment;
11. Has a undergone ocular surgery in the past 6 months;
12. Uses warm compress therapy, unless performed regularly, for a minimum of 30 days, and maintained at the same frequency throughout the duration of the study;
13. Unwilling to stop using their habitual ocular lubricants or artificial tears after Visit 2 (start of Part II);
14. Has been fitted with punctal plugs within 30 days prior to Screening;
15. Is a member of the Centre for Ocular Research & Education directly involved in the study;
16. Has taken part in another clinical research study within the last 30 days.

    * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 1 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 5 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 15 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 30 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 60 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 90 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness
Non-Invasive Tear Break Up Time "NITBUT" duration | Part I: 120 minutes after instillation
  NITBUT is measured in seconds. A NITBUT less than 10 seconds indicates eye dryness

SECONDARY OUTCOMES:
Tear Meniscus Height (TMH) Assessment | Part I: 5-15-30-60-90-120 minutes after instillation
  TMH assessment is measured in millimeters. TMH less than 0.2mm indicated eye dryness
Lipid Layer Thickness (LLT) Assessment | Part I: 5-15-30-60-90-120 minutes after instillation
  LLT is assessed in nanometer. A LLT less than 100nm indicates eye dryness
Ocular Surface Disease Index "OSDI" score | (Part II: after 7 days of consecutive I-DROP MGD usage)
  The OSDI is assessed on a scale of 0 and 100. A higher composite score indicates more severe eye dryness
Standard Patient Evaluation of Eye Dryness Score "SPEED questionnaire" | (Part II: after 7 days of consecutive I-DROP MGD usage)
  SPEED questionnaire is assessed on a scale from 0 to 28. A higher composite score indicates more severe eye dryness
Subjective measurement of "Change in comfort" | (Part II: At baseline and after 7 days of consecutive I-DROP MGD usage)
  Participants will rate their eye comfort on a 0-100 scale, where 0=poor comfort, 100=excellent comfort
Subjective measurement of "Change in Dryness" | (Part II: At baseline and after 7 days of consecutive I-DROP MGD usage)
  Participants will rate their eye dryness on a 0-100 scale, where 0=extremely dry, 100=no dryness
Subjective measurement of "Change in soothing" | (Part II: At baseline and after 7 days of consecutive I-DROP MGD usage)
  Participants will rate their experience of soothing on a 0-100 scale, where 0=no soothing, 100=extremely soothing
Subjective measurement of "Change in quality of vision" | (Part II: At baseline and after 7 days of consecutive I-DROP MGD usage)
  Participants will rate their quality of vision on a 0-100 scale, where 0=poor vision, 100=clear vision

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Ph.D., Principal Investigator — Centre for Ocular Research and Education
Locations (2):
- Canada (2):
  - Centre for Ocular Research & Education, Toronto, Ontario
  - Centre for Ocular Research & Education (CORE), Waterloo, Ontario